CLINICAL TRIAL: NCT01581970
Title: Potentiation of Cetuximab by Tregs Depletion With Metronomic Cyclophosphamide in Metastatic Squamous Cell Cancers of Head and Neck
Brief Title: Potentiation of Cetuximab by Tregs Depletion With CSA in Advanced Head & Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012LS002
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Head and Neck Cancer; Head and Neck Squamous Cell Carcinoma
Keywords: head and neck cancer; metastatic squamous cell cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck; Neoplasms, Squamous Cell | interventions — Cyclophosphamide; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cetuximab/low dose Cyclophosphamide (Experimental): Safety population as defined by all patients receiving at least one treatment with cyclophosphamide on Day 1.
  Interventions: Drug: Cyclophosphamide; Drug: Cetuximab

INTERVENTIONS:
Drug: Cyclophosphamide — Patients will be given oral cyclophosphamide 50 mg twice daily to be self-administered starting the first day of therapy with weekly cetuximab for 12 weeks or until disease progression.
  Other Names: Cytoxan
Drug: Cetuximab — The initial dose of cetuximab 400 mg/m^2 is administered over 120 minutes followed by weekly infusions of cetuximab 250 mg/m^2 intravenously (IV) over 60 minutes.
  Other Names: Erbitux

SUMMARY:
This is a feasibility study to assess the effectiveness of cetuximab when administered with low dose oral cyclophosphamide. Patients with metastatic squamous cell cancer of head and neck who have progressed on first line chemotherapy other than a cetuximab containing regimen will be treated with standard of care weekly cetuximab and twice daily low dose oral cyclophosphamide for 12 weeks.

DETAILED DESCRIPTION:
In this study, patients with head and neck squamous cell carcinoma (HNSCC) will be given low-dose cyclophosphamide in combination with standard of care cetuximab. Tumor biopsies will be collected before and six weeks after treatment for measurement of tumor infiltration by effector cells, including CD8+ T cells, natural killer (NK) cells, and monocytes. In addition, the proportion of Regulatory T Cells (Tregs) to effector cells will be measured in peripheral blood at the same time points.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented squamous cell carcinoma of the head and neck (irrespective of site of primary - nasopharyngeal, oral cavity, oropharyngeal, laryngeal or unknown primary) that is metastatic/incurable and has progressed on a first line chemotherapy regimen.
* Progression of measurable disease within the last 6 weeks based on Response Evaluation Criteria in Solid Tumors (RECIST) criteria
* If the patient has received prior treatment with anti-epidermal growth factor receptor (EGFR) therapy as a part of definitive therapy concurrent with radiation, the time from the last cetuximab exposure must be > 180 days.
* Must be at least 30 days from prior treatment and have recovered from the reversible effects of previous anti-cancer treatment
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0, 1 or 2
* Adequate bone marrow, renal and hepatic function within 14 days of study enrollment defined as:

  * Bone marrow: White blood cells (WBC) > 3,000/uL; absolute neutrophil count > 1,500/uL; platelets > 100,000/uL
  * Renal: creatinine ≤ 2.5 times the institutional upper limit of normal (ULN)
  * Hepatic: total bilirubin < 1.5 X institutional ULN; aspartate aminotransferase/alanine aminotransferase (AST[SGOT] and ALT[SGPT]) < 2.5 X institutional ULN
  * Albumin > 3.0 gm/dL
* Women of childbearing potential and fertile men must be willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study and for 60 days after the last dose of study drug.
* Voluntary written consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care

Exclusion Criteria:

* Pregnant or lactating - females of child bearing potential must have a negative pregnancy test within 14 days of study enrollment as cyclophosphamide is Pregnancy Category D
* History of another active primary invasive cancer within the previous 2 years, excluding non-melanoma skin cancer
* The patient is receiving concurrent treatment with other anticancer therapy, including chemotherapy, immunotherapy, hormonal therapy, radiotherapy (RT), chemoembolization, or targeted therapy. Patients receiving palliative radiation therapy to bony metastases prior to the first dose of study medication are eligible.
* Chronic steroid dependence
* Known HIV-positive patients and those with other acquired/inherited immunodeficiency hepatitis B, hepatitis C, connective tissue disease, or other clinical diagnosis, ongoing or intercurrent illness that in the Investigator's opinion should preclude the subject from participation
* History of gastrointestinal disease causing malabsorption or obstruction such as, but not limited to Crohn's disease, celiac sprue, tropical sprue, bacterial overgrowth/blind loop syndrome, gastric bypass surgery, strictures, adhesions, achalasia, bowel obstruction, or extensive small bowel resection
* Inability to take medications by mouth
* History of allergic reactions attributed to compounds of similar chemical or biologic composition
* Active autoimmune disease, chronic inflammatory condition, conditions requiring concurrent use of any systemic immunosuppressants or steroids. Mild-intermittent asthma requiring only occasional beta-agonist inhaler use or mild localized eczema will not be excluded.
* Previous allo-transplant of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Jha, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression
Description: The number of patients without disease progression two years out from study enrollment. Progression of disease is defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria and is as at least a 20% increase in size of the lesion(s) being followed and/or the appearance of one or more new lesions.
Time Frame: At 2 Years
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 7
Participants | 1

2. Secondary Outcome: Aggregate Ratio of Tregs to Effector Cells for All Participants
Description: The ratio of Tregs to effector cells (NK cells, CD 8+ lymphocytes, macrophages/monocytes) in tumor tissue as measured by immune-histochemistry (IHC) of tumor tissue for all Participants. Measure of central tendency was collected but the data is not accessible anymore because PI left institution and did not respond to requests for data.
Time Frame: 6 Weeks Post Treatment with Cyclophosphamide
Measure: Number; unit: ratio
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 4
ratio | 0.112

3. Secondary Outcome: Aggregate Ratio of Tregs to Natural Killer (NK) Cells for All Participants
Description: the Ratio of Tregs to NK cells in peripheral blood as measured by flow cytometry for all Participants. Measure of central tendency was collected but the data is not accessible anymore because the PI left institution and did not respond to requests for data.
Time Frame: 6 Weeks Post Treatment with Cyclophosphamide
Population: Measure of central tendency could not be used as the data was not originally reported in this manner and is not accessible anymore because the PI left institution and did not respond to requests for data.
Measure: Number; unit: ratio
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 4
ratio | 2.443

4. Secondary Outcome: Myeloid-derived Suppressor Cells in Tumor Tissue
Description: Myeloid-derived suppressor cells in tumor tissue as measured by immune-histochemistry (IHC)
Time Frame: Week 6
Population: This outcome measure was considered to not be helpful and the data was not collected.
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 0

5. Secondary Outcome: Quality of Life Scores
Description: Comparison of health related quality of life scores as measured by FACT-G: Functional Assessment of Cancer Therapy - General (constitutes the core of all subscales; the FACT-G can be used with patients of any tumor type)questionnaire.
  At this point, the data is not able to be analyzed because the PI left the institution and did not respond to requests for data.
Time Frame: Comparison from Baseline to Week 6 and Week 12
Population: At this point, the data is not able to be analyzed because the PI left the institution and did not respond to requests for data.
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 0

6. Secondary Outcome: Overall Survival
Description: Defined as the number of patients alive two years out from study enrollment.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Number analyzed (Participants) | 7
Participants | 1

ADVERSE EVENTS:
Arm/Group | Cetuximab/Low Dose Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab/Low Dose Cyclophosphamide (N=7)
Seizure (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab/Low Dose Cyclophosphamide (N=7)
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 2
Cerumen Impaction (Ear and labyrinth disorders) | 1
Fatigue (General disorders) | 2
Fever (General disorders) | 2
Odynophagia (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Intestinal Stoma Leak (Injury, poisoning and procedural complications) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Oral Pain (Gastrointestinal disorders) | 1
Neck Mass Pain (General disorders) | 1
Extremity Pain (Musculoskeletal and connective tissue disorders) | 1
Rash, Papulopustular (Skin and subcutaneous tissue disorders) | 1
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Rash, Maculopapular (Skin and subcutaneous tissue disorders) | 5
Rash, Acneiform (Skin and subcutaneous tissue disorders) | 1
Scalp Pain (Skin and subcutaneous tissue disorders) | 1
Skin Infection (Infections and infestations) | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Thromboembolic Event (Vascular disorders) | 1
Urinary Tract Infection (Infections and infestations) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No